CLINICAL TRIAL: NCT06096610
Title: The Effects of Resistance Training on Muscle Lipids in Children.
Brief Title: Resistance Training in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Strength and Conditioning Association (Other)
Responsible Party: Principal Investigator, Trent J. Herda, Ph.D., Professor, University of Kansas Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY0014990
Record Dates: First submitted 2023-10-17; First posted 2023-10-24 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Healthy
Keywords: exercise; muscle cross-sectional area; intramyocellular lipids; extramyocellular lipids; strength
MeSH Terms: conditions — Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Resistance exercise training (Experimental): Participants undergo 24 sessions of resistance exercise training over about 8 weeks.
  Interventions: Other: Resistance exercise training
- Control (No Intervention): Participants do not perform resistance exercise training.

INTERVENTIONS:
Other: Resistance exercise training — Participants will strength train via linear periodization resistance exercise training.
  Arms: Resistance exercise training

SUMMARY:
The project is going to examine the effects of resistance exercise training in prepubescent youth on skeletal muscle strength and lipid content.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer males and females ages 8 - 10 years.

Exclusion Criteria:

* No history or ongoing neuromuscular diseases.
* No history or ongoing musculoskeletal injuries.
* No history or ongoing disease that effects metabolism.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-10-14 (Actual); Study Completion 2023-10-14 (Actual)

PRIMARY OUTCOMES:
Change in the muscular strength of leg extensors, as measured with isotonic strength. | baseline, following the intervention (9 weeks)
  The score will reflect the strength of the leg extensors. The higher score, reflects greater muscular strength.

SECONDARY OUTCOMES:
Change from baseline in thigh muscle cross-sectional area. | baseline, following the intervention (9 weeks)
  Scores are measured cross-sectional area from ultrasound images. The higher score, reflects greater muscle size of the leg extensors.

OTHER OUTCOMES:
Change from baseline in intramyocellular lipids of the vastus lateralis, as measure with magnetic resonance spectroscopy | baseline, following the intervention (9 weeks)
  The score will reflect a concentration. The higher score, reflects more fat in the fibers.
Change from baseline in extramyocellular lipids of the vastus lateralis, as measure with magnetic resonance spectroscopy | baseline, following the intervention (9 weeks)
  The score will reflect a concentration. The higher score, reflects more fat in the fibers.
Change from baseline in the fatty acid saturation levels of the extramyocellular lipids of the vastus lateralis, as measure with magnetic resonance spectroscopy | baseline, following the intervention (9 weeks)
  The score will reflect a saturation level of fatty acids in the extramyocellular lipid. The higher score, reflects greater fatty acid saturation.
Change from baseline in the fatty acid saturation levels of the intramyocellular lipids of the vastus lateralis, as measure with magnetic resonance spectroscopy | baseline, following the intervention (9 weeks)
  The score will reflect a saturation level of fatty acids in the intramyocellular lipid. The higher score, reflects greater fatty acid saturation.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Hoglund Biomedical Imaging Center, Kansas City, Kansas
  - Exercise and Human Performance Laboratory, Overland Park, Kansas
  - Metabolic and Body Composition Laboratory, Overland Park, Kansas

IPD SHARING:
Plan to Share IPD: No